CLINICAL TRIAL: NCT04475757
Title: Effectiveness Of Ultra Sounded Guided Posterior Transverses Abdominis Plane & Lateral Femoral Cutaneous Nerve Blocks For Analgesia After Hip Hemiarthroplasty
Brief Title: Ultra Sounded Guided Posterior Transverse Abdominis Plane & Lateral FEMORAL Cutaneous Nerve Blocks Analgesia Post Hip Hemiarthroplasty
Status: Completed | Type: Observational
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Dr Manar Mamdouh Fahmy Elsharkawi, SPECIALIST ANESTHESIA, Dubai Health Authority
Other Study IDs: DSREC-02/2018_05
Record Dates: First submitted 2020-06-26; First posted 2020-07-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COMBINED ULTRASOUND GUIDED POSTERIOR TRANS VERSUS ABDOMINAL PLANE & LATERAL FEMORAL CUTANEOUS NERVE BLOCKS FOR POSTOPERATIVE ANALGESIA AFTER HIP HEMIARTHROPLASTIC SURGERY

DETAILED DESCRIPTION:
TO EVALUATE THE EFFECTIVENESS OF POSTOPERATIVE ANALGESIA FOR HIP HEMIARTHROPLASTIC SURGERIES BY USING ULTRASOUND GUIDED POSTERIOR TRANS VERSUS ABDOMINAL PLANE & LATERAL FEMORAL CUTANEOUS NERVE BLOCKS

ELIGIBILITY:
Inclusion Criteria:

* Hemiarthroplaty surgery
* ASA 1 - ASA 4

Exclusion Criteria:

* ALLERGIC TO LOCAL ANESTHETICS
* PATIENT REFUSAL

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: POSTOPERATIVE PATIENT UNDERGOING HIP HEMIARTHROPLASTIC SURGERY
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
PAIN MANAGEMENT | 2 DAYS
  POSTOPERATIVE ANALGESIA

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Health Authority, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No